CLINICAL TRIAL: NCT03270150
Title: Evaluation of Safety and Efficacy of the BTL-899 Device for Non-invasive Lipolysis and Circumference Reduction of Abdomen
Brief Title: Effect of the BTL-899 Therapy for Non-invasive Lipolysis and Circumference Reduction of Abdomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899L
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Improvement of Abdomen Appearance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BTL-899 Therapy Arm (Experimental): BTL-899 therapy, 3 therapies
  Interventions: Device: BTL-899

INTERVENTIONS:
Device: BTL-899 — BTL-899

SUMMARY:
The study is a prospective open-label single-arm study that includes three treatment procedures and four follow-up visits.

DETAILED DESCRIPTION:
This study will evaluate the clinical efficacy and safety of the BTL-899 device for non-invasive lipolysis and circumference reduction of abdomen. The study is a prospective open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will complete three (3) treatment visits and will be invited to four (4) follow-up visits 1, 2, 3 and 6-months after the final treatment. 6-months follow-up visit is the optional one.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Voluntarily signed informed consent form
* BMI ≤ 35 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Cardiac pacemakers
* Cardiovascular diseases
* Implanted defibrillators, implanted neurostimulators
* Electronic implants
* Disturbance of temperature or pain perception
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Malignant tumor
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contageous skin disease
* Elevated body temperature
* Pregnancy
* Breastfeeding
* Injured or otherwise impaired muscles
* Scars, open lesions and wounds at the treatment area
* Basedow's disease
* Previous liposuction in the treatment area in the last six months
* Abdominal wall diastasis
* Unstable weight within the last 6 months
* Previous body contouring treatments in the abdomen area in the last three months

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of the BTL-899 treatment for abdomen circumference reduction after the final follow-up visit | 4 months
  Evaluation of change in abdomen circumference using tape measurements in cm at the final follow-up visit.
Occurrence of adverse events | 7 months
  The occurrence of adverse events will be followed throughout the whole study.

SECONDARY OUTCOMES:
Efficacy of BTL-899 treatment for fat and circumference reduction in abdomen, as assessed by two blinded evaluators | 4 months
  Evaluation of photographs before and after the treatment.
Efficacy of the BTL-899 treatment for abdomen circumference reduction | 4 months
  Evaluation of change in abdomen circumference using tape measurements in cm at all study visits after the first therapy.
Ultrasound imaging | 4 months
  Evaluation of ultrasound images.
Subject's satisfaction with study treatment | 4 months
  Subject's satisfaction with the therapy results evaluated through the Subject Satisfaction Questionnaire (5-point scale).
Therapy comfort during the study treatment. | 1 month
  Therapy comfort during the treatment evaluated through the Therapy Comfort Questionnaire (10-point scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Aesthe Clinic, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No